CLINICAL TRIAL: NCT03968263
Title: The Effects of Different Activation Protocols of Hycon Device and Vibration Stimulation on Orthodontic Canine Teeth Distalization
Brief Title: The Effects of Different Activation Protocols of Hycon Device and Vibration Stimulation on Canine Teeth Distalization
Acronym: Acceleration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ahmet Yağcı, Associate Professor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TDH-2019-8701; TDH-2019-8701 (Other Grant/Funding Number: Republic Of Turkey, Erciyes University)
Record Dates: First submitted 2019-04-12; First posted 2019-05-30 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Tooth Migration
Keywords: Vibration; Tooth movement acceleration
MeSH Terms: conditions — Tooth Migration

STUDY DESIGN:
Intervention Model Description: Routine orthodontic treatment procedures will be applied to patients
Who Masked: Participant, Outcomes Assessor
Masking Description: It will not be possible to prevent clinicians and their interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Hycon device(Routine protocol) (Active Comparator): The hycon device in this group will be activeted into half turn every 3 days in accordance with the manufacturer's instructions.
  Interventions: Device: Hycon device(Routine protocol); Device: Hycon device(Modified protocol); Device: Hycon device(Routine protocol) and Vibration(Acceledent); Device: Hycon device(Modified protocol) and Vibration(Acceledent)
- Hycon device(Modified protocol) (Active Comparator): The activation period of the hycon device in this group will be modified. The first day will be clockwise half a turn, the second day will be half-turn clockwise and the third day will be turned half a turn counterclockwise.
  Interventions: Device: Hycon device(Routine protocol); Device: Hycon device(Modified protocol); Device: Hycon device(Routine protocol) and Vibration(Acceledent); Device: Hycon device(Modified protocol) and Vibration(Acceledent)
- Hycon device(Routine protocol) and Vibration (Active Comparator): The hycon device in this group will be activeted into half turn every 3 days in accordance with the manufacturer's instructions. In addition, patients in this group twice a day for 10 minutes with acceledent device vibration will be applied.
  Interventions: Device: Hycon device(Routine protocol); Device: Hycon device(Modified protocol); Device: Hycon device(Routine protocol) and Vibration(Acceledent); Device: Hycon device(Modified protocol) and Vibration(Acceledent)
- Hycon device(Modified protocol) and Vibration (Active Comparator): The activation period of the hycon device in this group will be modified. The first day will be clockwise half a turn, the second day will be half-turn clockwise and the third day will be turned half a turn counterclockwise. In addition, patients in this group twice a day for 10 minutes with acceledent device vibration will be applied.
  Interventions: Device: Hycon device(Routine protocol); Device: Hycon device(Modified protocol); Device: Hycon device(Routine protocol) and Vibration(Acceledent); Device: Hycon device(Modified protocol) and Vibration(Acceledent)

INTERVENTIONS:
Device: Hycon device(Routine protocol) — Hycon device will be activated half a turn every 3 days.
Device: Hycon device(Modified protocol) — The activation period of the hycon device will be modified.
Device: Hycon device(Routine protocol) and Vibration(Acceledent) — Hycon device will be activated half a turn every 3 days. Vibration will be applied 2 times 10 minutes per day.
Device: Hycon device(Modified protocol) and Vibration(Acceledent) — The activation period of the hycon device will be modified. Vibration will be applied 2 times 10 minutes per day.

SUMMARY:
This study will be performed with 25 patients who applied to Erciyes University Faculty of Dentistry for treatment and who need 2 first premolar extraction and maximum anchorage for treatment. In order to increase anchorage in the patient who will start the distalization of canine, mini screw (1.5 mm diameter, 7 mm length) will be applied to the right and left maxillary dentition of the patient under local anesthesia. The hycon device, which has a screw-shaped design for the application of force to both the right and left sides of the maxillary dentition of the patients, will be adapted to the bands in the 1st molar teeth. Patients will be randomly divided into 4 groups. Vibration will be applied to the two groups with the Acceledent device.

Group 1 = The hycon device in this group will be used in accordance with the manufacturer's instructions.

Group 2 = The activation period of the hycon device in this group will be modified.

Group 3 = The hycon device in this group will be used in accordance with the manufacturer's instructions. In addition, patients in this group twice a day for 10 minutes with acceledent device vibration will be applied.

Group 4 = The activation period of the hycon device in this group will be modified. In addition, patients in this group twice a day for 10 minutes with acceledent device vibration will be applied.

The period of canine distalization of orthodontic treatment is one of the important stages affecting the duration of treatment. Shortening this time in the clinic will shorten the duration of treatment.

If this application changes the tooth movement speed in any direction, it will support the new research.

DETAILED DESCRIPTION:
This study is planned as a splint mouth, randomized, non-controlled clinical trial.This study will be performed with 25 patients who applied to Erciyes University Faculty of Dentistry for treatment and who need 2 first premolar extraction and maximum anchorage for treatment.Patients will be selected from 12 to 18 years of age.In order to increase anchorage in the patient who will start the distalization of canine, mini screw (PSM Medical Solutions, Quattro Standard Screw 1,5x7mm, Tuttlingen,Germany) will be applied to the right and left maxillary dentition of the patient under local anesthesia.The hycon device (Adenta,Germany), which has a screw-shaped design for the application of force to both the right and left sides of the maxillary dentition of the patients, will be adapted to the bands in the 1st molar teeth.The approval of the study was taken from Erciyes University Clinical Research Ethics Committee in Kayseri (2018/337).Informed consent will be obtained from all patients included in the study.Consent will be taken from parents of those under the age of 18. At the beginning of the treatment and at the end of the treatment, all patients who participated in the study received standard treatment records including photographs, dental models and radiography.

Inclusion criteria:

* No systemic disease
* Being healthy as periodontal.
* No smoking.
* No previous orthodontic treatment.
* Lack of congenital tooth deficiency
* Permanent dentition
* Indication of extraction for 1.premolar in the maxilla
* There is no restoration of upper canine teeth.
* Indication of the use of mini screw for maximum anchoring in the maxilla

All models will be scanned by 3D laser model scanning device (3 Shape, R 700 Desktop Scanner, Szczecin, Poland) and digitalized (3Shape Ortho Analyzer ™ 12). The gradient of the teeth and the amount of space closure will be examined by using panoramic radiographs. The amount of root resorption in canine teeth will be measured by using periapical radiography. As a result of the data obtained, the effects of the hycon device(Adenta, Germany) and vibration device(Acceledent Aura, OrthoAccel Technologies, Inc. USA) on the tooth movement speed will be compared.

ELIGIBILITY:
Inclusion Criteria:

* No systemic disease
* Being healthy as periodontal.
* No smoking.
* No previous orthodontic treatment.
* Lack of congenital tooth deficiency
* Permanent dentition
* Indication of extraction for 1.premolar in the maxilla
* There is no restoration of upper canine teeth.
* Indication of the use of mini screw for maximum anchoring in the maxilla

Exclusion Criteria:

* Orthodontic treatment history
* Missing tooth
* Poor oral hygiene
* Lack of cooperation

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-02-08 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2021-02-08 (Estimated)

PRIMARY OUTCOMES:
Acceleration of tooth movement | 2 year
  maxillary canine distal movement amount (mm)

SECONDARY OUTCOMES:
Reduction of pain during treatment | 2 year
  measurement of pain level (grading system, VAS scoring)
Shortening of total treatment time | 2 year
  measurement of treatment time (months)

CONTACTS AND LOCATIONS:
Overall Officials: Osman Yildiz, Research as., Study Chair — Research as.
Locations (1):
- Erciyes University, Faculty of Dentistry, Department of Orthodontics University university, Kayseri, Melikgazi, Turkey (Türkiye)

REFERENCES:
- [Background] McLaughlin RP, Kalha AS, Schuetz W. An alternative method of space closure: the Hycon Device. J Clin Orthod. 2005 Aug;39(8):474-84; quiz 471. No abstract available. PMID 16247198
- [Background] Elmotaleb MAA, Elnamrawy MM, Sharaby F, Elbeialy AR, ElDakroury A. Effectiveness of using a Vibrating Device in Accelerating Orthodontic Tooth Movement: A Systematic Review and Meta-Analysis. J Int Soc Prev Community Dent. 2019 Jan-Feb;9(1):5-12. doi: 10.4103/jispcd.JISPCD_311_18. Epub 2019 Feb 14. PMID 30923687
- See also: pubmed ID not found — https://progressinorthodontics.springeropen.com/articles/10.1186/2196-1042-14-42